CLINICAL TRIAL: NCT01830933
Title: Breast Cancer Risk Reduction: A Patient Doctor Intervention
Acronym: BreastCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); California Breast Cancer Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 150B-0158; NCT01836250 (obsolete NCT alias)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer concern, breast cancer risk perception, breast cancer risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BreastCARE Intervention (Experimental): Intervention Clinic Patients: The RA will welcome the patient upon arrival at the clinic and again explain study procedures and field any questions. The RA will have the patient sign the HIPAA authorization form and then demonstrate how to enter information and answer questions on the tablet-PC and the patient will indicate their consent electronically before beginning the assessment.
  Intervention Patient Report. Once the patient completes the BreastCare Computer survey, the program will immediately generate a personal feedback report containing information about her risk factors and recommendations to reduce her risk. This report will be printed and given to the patietns before she meets with her doctor.
  Interventions: Other: BreastCARE
- BreastCARE Comparison (No Intervention): Patients will be randomized into the intervention or comparison groups at the time of recruitment. Block-randomization will be used to assign patients to intervention or comparison groups.
  Comparison Clinic Patients. Contact and baseline interview procedures will be the same for patients from the comparison clinics, however there will be no computer assessment at the time of their clinic visit. An RA will meet the patient 10 minutes prior to her appointment time to obtain written HIPAA authorization.

INTERVENTIONS:
Other: BreastCARE — Physician Report. At the time of an individual participant's visit to her primary care physician and her completion of the assessment tool, her physician will receive a physician report. The physician report is designed to facilitate communication about breast cancer risk during the primary care visit and to provide tailored risk reduction recommendations.
  Arms: BreastCARE Intervention

SUMMARY:
The proposed research combines the scientific advances in breast cancer research with health information technology (IT) to design a personalized intervention that assesses breast cancer risk for women, disseminates important breast health information, and facilitates discussion of breast cancer risk reduction practices. Our goal is to implement a tablet-PC (personal computer) based breast cancer risk education (BreastCare) intervention in the primary care setting that estimates a woman's individual risk for breast cancer and provides her and her physician with personalized breast cancer risk information and recommendations for action.

ELIGIBILITY:
Inclusion Criteria:

1. Patient component:

   * Women who visit the General Internal Medicine (GIM) practices at SFGH and UCSF during the study period
   * Between the ages of 40 and 74
   * Self-identify as Asian American, Spanish- and English-speaking Latinas, African American, or White
   * Have no history of breast cancer are eligible to participate.
2. Physician component: Primary care physicians currently practicing at the GIM clinics at SFGH and UCSF

Exclusion Criteria:

1. Patient component: Women whose physicians object to their participation in the study
2. Physician component: No exclusion criteria for physicians

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1235 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celia P Kaplan, DrPH, MA, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital (SFGH), San Francisco, California
  - University of California, San Francisco Mt. Zion campus, San Francisco, California

REFERENCES:
- [Derived] Livaudais-Toman J, Karliner LS, Tice JA, Kerlikowske K, Gregorich S, Perez-Stable EJ, Pasick RJ, Chen A, Quinn J, Kaplan CP. Impact of a primary care based intervention on breast cancer knowledge, risk perception and concern: A randomized, controlled trial. Breast. 2015 Dec;24(6):758-66. doi: 10.1016/j.breast.2015.09.009. Epub 2015 Oct 21. PMID 26476466

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual Care is the comparison Clinic Patients, where there is no change in their standard or usual care.
- BreastCARE Intervention: Intervention Clinic Patients: The participants will answer questions on the tablet-PC to calculate their breast cancer risk.
  Intervention Patient Report. Once the patient completes the BreastCare Computer survey, the program will immediately generate a personal feedback report containing information about her risk factors and recommendations to reduce her risk. This report will be printed and given to the patients before she meets with her doctor.
  BreastCARE : The physician will receive a physician report that contains information similar to the patient report.
Period: Overall Study
Arm/Group | Usual Care | BreastCARE Intervention
Started | 823 | 812
Completed Meet-up | 675 | 603
Completed | 655 | 580
Not Completed | 168 | 232

BASELINE CHARACTERISTICS:
Population: Number of participants who completed follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | BreastCARE Intervention | Total
Number analyzed (Participants) | 655 | 580 | 1235
Age, Customized [Number; unit: participants]
  <50 years | 183 | 182 | 365
  51-65 years | 362 | 300 | 662
  >65 years | 110 | 98 | 208
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 655 | 580 | 1235
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Latina White | 229 | 202 | 431
  Latina | 144 | 141 | 285
  Black/ African American | 150 | 125 | 275
  Asian or Pacific Islander | 123 | 105 | 228
  Native American or Other | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 655 | 580 | 1235

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Breast Cancer Risk Factors
Description: Risk knowledge was assessed using a post-survey. Participants could have scored 0-100 (with 0 meaning no correct answers, and 100 is all correct answers). This outcome was measured through a survey. Breast cancer risk knowledge was based on a series of eight questions in the survey. O
Time Frame: one week post-initial visit (approximately one week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | BreastCARE Intervention
Number analyzed (Participants) | 655 | 580
units on a scale | 48.9 (24.3) | 56.4 (24.3)

2. Primary Outcome: Percentage of Participants With Correct Perception of Risk
Description: This outcome was measured through a survey. Women were asked what they thought about their risk of getting breast cancer was compared to other women of the same age.
Time Frame: baseline, one week post-initial visit (approximately one week)
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | BreastCARE Intervention
Number analyzed (Participants) | 655 | 580
percentage of participants
  Baseline | 69.9 | 65.9
  Final (one week post-intial visit) | 73.3 | 71.1

3. Primary Outcome: Percentage of Participants Who Had a Discussion of Breast Cancer Risk
Description: Self-reported discussion of breast cancer risk with physicians.
Time Frame: one week post-initial visit (approximately one week)
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | BreastCARE Intervention
Number analyzed (Participants) | 655 | 580
percentage of participants | 15 | 41

4. Primary Outcome: Percentage of Participants Who Reported Discussion of Mammography Screening
Description: Self reported discussion of mammography with physician.
Time Frame: up to 14 months
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | BreastCARE Intervention
Number analyzed (Participants) | 655 | 580
percentage of participants | 51.6 | 61.5

ADVERSE EVENTS:
Arm/Group | Usual Care | BreastCARE Intervention
Serious Adverse Events (participants affected / at risk) | 0/655 | 0/580
Other Adverse Events (participants affected / at risk) | 0/655 | 0/580

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No